CLINICAL TRIAL: NCT06906146
Title: Effectivness of Capacitive Resistive Electric Transfer Therapy on Muscle Recovery in Athletes
Brief Title: Capacitive Resistive Electric Transfer Therapy on Muscle Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CBAS-2023-03
Record Dates: First submitted 2025-03-06; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Muscle Oxygenation; Lactate; Anaerobic Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CRET therapy (Experimental)
  Interventions: Device: CRET therapy
- Sham (Sham Comparator)
  Interventions: Device: Sham CRET Therapy

INTERVENTIONS:
Device: CRET therapy — Capacitive Resistive Electric Transfer (CRET) therapy is a treatment modality that applies high-frequency electrical currents to stimulate tissue regeneration, enhance blood circulation, and reduce muscle pain. It operates through two modes: the capacitive mode, which targets superficial tissues such as skin and muscle, and the resistive mode, which penetrates deeper structures like tendons, ligaments, and joints. This technique is widely used in rehabilitation, sports physiotherapy, and pain management to accelerate muscle recovery and optimize neuromuscular function.
  Arms: CRET therapy
Device: Sham CRET Therapy — Same as CRET therapy but in a aham form.
  Arms: Sham

SUMMARY:
This study aims to evaluate the effectiveness of Capacitive Resistive Electric Transfer (CRET) therapy combined with post-competition massage in the recovery and muscle function of professional athletes. It is designed as a randomized, double-blind, crossover clinical trial. The primary objective is to analyze the efficacy of this combined protocol in muscle recovery after performing the Wingate anaerobic power and capacity test. Secondary objectives include assessing changes in muscle fatigue, muscle function of the rectus femoris and vastus lateralis, physiological changes in blood lactate concentration and oxygen saturation, and intramuscular structural changes through ultrasound before and after the intervention.

The study will recruit professional athletes from disciplines that require anaerobic muscle metabolism, such as cycling, athletics, triathlon, CrossFit, and duathlon. Participants must be federated athletes who train at least four times per week and actively compete at regional, national, or international levels. Exclusion criteria include recent sports injuries preventing test performance, prior exposure to CRET therapy, allergies to conductive gel, language barriers, participation in other research studies, or ongoing pharmacological treatment that could interfere with measurements.

Participants will attend four study sessions, divided into two sets of two consecutive days. On the first day, they will perform the Wingate test followed by the assigned post-competition massage with either CRET therapy or a placebo intervention. On the second day, they will repeat the Wingate test. After a three-week washout period, participants will switch to the opposite group. The intervention group will receive a 60-minute CRET therapy session with both resistive and capacitive modes applied at different power intensities, combined with a standardized recovery massage. The placebo group will receive the same massage while undergoing a simulated CRET therapy, with the machine turned on but without power application to prevent participant awareness of the placebo condition.

The study will analyze various dependent variables, including Wingate test performance, blood lactate levels, subjective fatigue perception using the modified Borg scale, muscle stiffness and tone through myotonometry, muscle oxygen saturation via near-infrared spectroscopy (NIRS), cross-sectional muscle area and grayscale values from ultrasound imaging, body composition using a Tanita analyzer, maximum isometric quadriceps strength via handheld dynamometry, and muscle activity measured by surface electromyography (sEMG). Each of these variables will be assessed at specific time points before, during, and after the intervention.

The estimated sample size is approximately 50 subjects, with 25 participants per group, determined through a preliminary pilot study. Statistical analyses will be conducted using IBM SPSS Statistics 26.0. Descriptive statistics will be calculated for quantitative and qualitative variables. A linear mixed model will be applied to compare changes between and within groups over five measurement periods using a one-way mixed ANOVA. If the sphericity assumption is violated, the Greenhouse-Geisser correction will be applied. Statistically significant effects will undergo post-hoc analysis with Bonferroni correction for multiple comparisons. All originally enrolled participants will be included in the final analysis following an intention-to-treat approach, and effect sizes will be calculated using eta squared. The significance level will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Athletes who practice a type of sport that requires the use of anaerobic muscle metabolism (cycling, athletics, triathlon, crossfit, spinning and duathlon)
* Athletes must be federated and train a minimum of 4 days/week
* Active participation in regional, national or international competitions.

Exclusion Criteria:

* Volunteers who have suffered a sports injury that makes it impossible for them to perform the test
* Having received the CRET therapy technique.
* Subjects who report allergies to the conductive cream.
* Subjects undergoing pharmacological medical treatment that may interfere with the measurements.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Lactate | 1 hour after the test
  Capacitive resistive electrical transfer therapy (CRET) is a treatment modality that applies high-frequency electrical currents to stimulate tissue regeneration, improve blood circulation and reduce muscle pain. It works through two modes: the capacitive mode, which targets superficial tissues such as skin and muscle, and the resistive mode, which penetrates deeper structures such as tendons, ligaments and joints. This technique is widely used in rehabilitation, sports physiotherapy and pain management to accelerate muscle recovery and optimize neuromuscular function.

SECONDARY OUTCOMES:
Wingate Test | During the test
  The Wingate test is used to determine power and anaerobic capacity (21). Each subject will perform the test: 30 seconds at maximum intensity interspersed with 1 minute of active recovery (pedaling 100 rpm), and this cycle will be repeated 3 times. The cycloergometer (Monark 818E, Vansbro, Sweden) will be used.
  The test will be performed with a flywheel load resistance calculated based on 0.075 kg of the subject's current body weight. Heart rate during the test will be monitored with a heart rate monitor (Polar CS100 Cycling Heart Rate Monitor).
Muscle oxygen saturation percentage | During the test
  Near infrared spectroscopy (NIRS) monitoring detects changes in tissue oxygenation in small blood vessels, capillaries and oxygen transport (e.g. myoglobin). This instrument determines the relationship between oxyhemoglobin concentration and total hemoglobin concentration in the muscle. The sensors will be attached to the vastus lateralis and rectus femoris muscles during the Wingate test.
Muscle thickness | 1 hour after the test
  Ultrasound (US) images were used (US Aloka Prosound C3 15.4) with a high-frequency linear transducer (USTTL01, 12 L5), measured by a researcher with more than 10 years of experience handling the instrument. Measurements were taken in the muscle belly of the vastus lateralis (i.e., in the same location as the NIRS measurements) and the rectus femoris, with the patient lying on the examination table, knees fully extended, and legs without rotation. Ultrasound imaging was always performed at the same point (marked with a dermographic pen), with the linear transducer placed at the same angle (perpendicular to the skin). The 90º angulation of the transducer was verified before each measurement using a goniometer. The transducer was positioned without applying force to the skin, merely making contact with the ultrasound gel. Ultrasound device settings were adjusted for each patient to optimize the visualization of the target tissue, and the same settings were maintained for all measurements
Maximal voluntary knee extension force | Before the test
  before (at rest) and the day after (24h after the end of the Wingate test and recovery intervention), subject performed a 5s isometric maximal voluntary contraction to measure the maximal voluntary force of the knee extensor muscles. The force was registered in the dominant lower limb and the unit of measure was Newtons. A traction dynamometer (PCE Ibérica S.L., Albacete, Spain) was used. During the assessment, participants were seated with their hips and knees flexed at a 90o angle, and a strap was secured on the distal and anterior part of the dominant leg. The test was repeated three times, and the mean value was used for the analysis. Verbal encouragements were given throughout the contraction time.
muscle activity | Before the test
  muscle activity was recorded using surface electromyography from vastus lateralis and rectus femoris. The data was obtained by consists of three parts: (a) a Shimmer3 sEMG unit (Realtime Technologies Ltd., Dublin, Ireland). The signal was smoothed using a window size of 0.025s root mean square (RMS) and an overlapping of 0.0125s between windows. The Maximal Voluntary Isometric Contraction (MVIC) was calculated using the peak of the RMS signal during the extension knee isometric test. The RMS was the principal variable recorded for muscle activity. The participants' skin was cleaned with alcohol and dried before the electrodes were placed. If hair impeded the correct adhesion of the electrodes to the skin, the particular site was shaved. Self-adhesive 5×5 cm Valutrode® surface electrodes were placed on the muscle bellies according to the SENIAM project recommendations and with an interelectrode distance of 20 mm. Vastus lateralis electrodes were placed between the line from

IPD SHARING:
Plan to Share IPD: No